CLINICAL TRIAL: NCT03827096
Title: Utilization of Autologous Mesenchymal Cells in Posterolateral Spinal Fusion in Degenerative Spine Disease to Assess the Safety and the Efficacy
Brief Title: Utilization of Autologous Mesenchymal Cells in Posterolateral Spinal Fusion in Degenerative Spine Disease
Acronym: AMSC-DSD-001
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Primary endpoint (Safety) has been achieved
Sponsor: Bioinova, s.r.o. (Industry)
Collaborators: University Hospital, Motol (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMSC-DSD-001
Record Dates: First submitted 2019-01-14; First posted 2019-02-01 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human AMSC (passage 3) 3P in 1.5 mL (Experimental): Patient receiving the investigational medicinal product - suspension of human autologous MSC 3P in 1.5 mL
  Interventions: Drug: Suspension of human autologous MSC 3P in 1.5 ml

INTERVENTIONS:
Drug: Suspension of human autologous MSC 3P in 1.5 ml — During the posterolateral spine fusion operation, 1.5 ml of cell suspension was mixed with 5cc of beta-tricalcium phosphate foam and 3.5 ml of patient's blood, and inserted between the right transverse processes of the lumbar spine.
  Other Names: hAMSC

SUMMARY:
Subjects in whom a posterolateral fusion surgery has been planned and who meet the inclusion and exclusion criteria were proposed to receive a single-dose AMSC treatment, in order to assess its safety and efficacy on posterolateral interbody fusion. After the surgery, the subjects were followed up as out-patients during 5 study visits for 12 months in total.

DETAILED DESCRIPTION:
Following informed consent collection at the screening visit and verification of all inclusion and exclusion criteria, eligible patients will undergo the procedure of bone marrow cell aspiration from iliac crest for the purpose of receiving autologous multipotent mesenchymal stem cells. The cells will be cultivated for 3 passages (for 3 - 4 weeks) in order to expand them to sufficient quantity. Suspension of the cultured AMSC will then be sterilely packed and transported to the surgery site. During the posterolateral spine fusion operation, 1.5 ml of cell suspension will be mixed with 5 cc of beta-tricalcium phosphate foam (Vitoss™, Orthovita) and 3.5 ml of patient's blood, and inserted between the transverse processes of the lumbar spine.

All subjects will be hospitalized and followed up as per standard medical care rules used in the investigational site hospital for this type of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. established diagnosis of spinal degenerative disease indicated for lumbar spine surgery,
2. patients indicated for fusion therapy,
3. patients between 18-55 years, both sexes,
4. patients able to provide written informed consent.

Exclusion Criteria:

1. previous lumbar spine surgery in the same segment of the spine, in order to achieve vertebral fusion,
2. osteoporosis,
3. diabetes mellitus,
4. pregnancy or breastfeeding,
5. women of childbearing potential not using effective contraception (established oral contraception, intrauterine device, ligation of the uterine tube) including proven contraceptive measures taken by their sexual partners,
6. fertile men not using proven contraceptive measures including effective contraception method in their partner (established oral contraception, intrauterine device, ligation of the uterine tube),
7. coagulopathy,
8. malnutrition, primary biliary cirrhosis,
9. skin infection at the site of bone marrow aspiration or at the site of spinal fusion,
10. gastrostomy,
11. any significant medical condition that would compromise the safety of the patient (e.g. recent myocardial infarction, congestive heart failure, renal failure, liver failure, systemic infection, recurrent thromboembolic disease .....),
12. alcohol or drug abuse,
13. cancer (compulsory clinical oncological screening),
14. ongoing or recent (last 3 months) systemic corticosteroid or immunosuppressive therapy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
Safety: To demonstrate absence of complications at the site of spinal fusion | 1 year
  Complications at the site of spinal fusion and other treatment-related adverse events will be recorded in ten patients at Visits I through VII. All adverse events (AEs) will be classified by seriousness, severity and relationship to hAMSC application.
  All AEs will be collected as symptoms spontaneously reported by the patient, clinically relevant changes and abnormalities observed by the Investigator (clinically significant laboratory measurements confirmed by repeated measurement, results of physical examinations) Intensity
  The following 3-point rating scale will be used for rating of the intensity of each AE:
  Mild: Awareness of signs or symptoms, but no disruption of usual activity Moderate: Event sufficient to affect usual activities (disturbing) Severe: Inability to work or perform usual activities (unacceptable)

SECONDARY OUTCOMES:
Efficacy: To assess the quality of life determined by Oswestry Questionnaire. | 1 year
  The quality of life determined by Oswestry Questionnaire will be recorded in ten patients at Visits II, and IV through VII. The test has 10 sections and maximum score is 50 points; change from the baseline valie will be recorded. The points are then transferred into percentage and interpreted in a standard way when 0-20% means minimal disability while 81-100% means bed-bound condition. Minimum detectable change (90 % confidence) is 10 % (5 points).
Efficacy: To assess the quality of spinal fusion by X-ray imaging | 1 year
  The quality of spinal fusion will be measured by X-ray imaging at Visits V and VII. Dynamic X-ray of the lumbar spine will be performed at 3 and 12 months following the surgery and hAMSC application to measure the angle of the spine movement in the fusion area. The angle will be recorded in degrees. The movements above 10 degrees will beregarded as "unstable".
  The bone fusion morphology will be evaluated based on the following scale:
  1. Cyst or pseudo-cyst formation
  2. Fusion not visible
  3. Pseudo-joint (or false joint) development
  4. Low degree of bone fusion
  5. High degree of bone fusion
Efficacy: To assess the quality of spinal fusion measured by computed tomography (CT). | 1 year
  The quality of spinal fusion will be measured by CT in ten patients at Visits V and VII.
  The density will of the fusion will be expressed as % on a linear scale between two standardized measuring points: soft tissue= 0%, vertebral arch= 100%.

IPD SHARING:
Plan to Share IPD: No
The data will be published